CLINICAL TRIAL: NCT01750853
Title: A Study of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of LY3045697 After Single Oral Dosing in Healthy Subjects
Brief Title: A Study of LY3045697 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 15035; I6S-MC-ASEA (Other: Eli Lilly and Company); 2012-004968-22 (EudraCT Number)
Record Dates: First submitted 2012-12-13; First posted 2012-12-17 (Estimated); Last update posted 2013-07-26 (Estimated); Status verified 2013-07

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Experimental): Period 1: 0.1 milligrams (mg) LY3045697 administered once orally or matching placebo administered once orally.
  Period 2: 1 mg LY3045697 administered once orally or matching placebo administered once orally.
  Period 3: 10 mg LY3045697 administered once orally or matching placebo administered once orally.
  Interventions: Drug: LY3045697; Drug: Placebo
- Group 2 (Experimental): Period 1: 0.3 mg LY3045697 administered once orally or matching placebo administered once orally.
  Period 2: 3 mg LY3045697 administered once orally or matching placebo administered once orally.
  Period 3: 30 mg LY3045697 administered once orally or matching placebo administered once orally.
  Interventions: Drug: LY3045697; Drug: Placebo
- Group 3 (Experimental): Period 1: 100 mg of LY3045697 administered once orally or matching placebo administered once orally.
  Period 2: 300 mg of LY3045697 administered once orally or matching placebo administered once orally (via split delivery over a 15-minute period).
  Interventions: Drug: LY3045697; Drug: Placebo

INTERVENTIONS:
Drug: LY3045697 — Administered orally
Drug: Placebo — Administered orally

SUMMARY:
The purpose of this study is to investigate the safety and tolerability of LY3045697 after a single dose, and to determine how long LY3045697 remains in the body. Two cohorts (groups) of 9 participants each will participate in 3 dosing periods. These participants will receive placebo in one period only. A third cohort of 9 will participate in 2 dosing periods and participants will receive either 2 dose levels of LY3045697 or 1 dose level of LY3045697 and placebo by the end of both periods.

DETAILED DESCRIPTION:
Cohort 3 added per protocol amendment (April, 2013).

ELIGIBILITY:
Inclusion Criteria:

* Are healthy males or females of non-child bearing potential as determined by medical history and physical examination
* Male participants must agree to use a medically accepted method of contraception with all sexual partners during the study and for 90 days after the end of the final dosing
* Female participants must be postmenopausal or surgically sterile
* Postmenopausal female participants are between the ages of 45 and 65 years, inclusive and must be 12 months without a menstrual period or 6-12 months without a menstrual period and Follicle-Stimulating Hormone (FSH) greater than (>) 40 International Units per Liter (IU/L)
* Have a body mass index (BMI) between 18.0 and 32.5 kilogram per square meter (kg/m²), inclusive, at entry
* Have clinical laboratory test results within normal reference range for the population or investigator site or results with acceptable deviations that are judged to be not clinically significant by the Medical Investigator (MI)
* Have venous access sufficient to allow blood sampling
* Are non-smokers or smoker of 5 or less cigarettes/cigars/pipes per day as determined by history
* Have the ability and willingness to abstain from alcohol, methylxanthine-containing beverages or food (coffee, tea, cola, chocolate, "power drinks"), poppy seed, and tobacco products from 48 hours prior to entry in the clinical research center until discharge

Exclusion Criteria:

* Are currently enrolled in, or discontinued within the last 60 days prior to drug administration inclusive from a clinical trial involving an investigational drug that has not received regulatory approval for any indication
* Have previously completed or withdrawn from this study or any other study investigating this study drug
* Have a history or presence of medical illness including but not limited to any cardiovascular, hepatic, respiratory, hematological, endocrine, psychiatric or neurological disease, or any clinically significant laboratory abnormality, that in the judgment of the MI, indicates a medical problem that would preclude study participation
* Have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the MI, increases the risks associated with participating in the study. In addition, participants with the following findings will be excluded:
* Confirmed corrected QT (QTcF) interval > 450 milliseconds (msec) for males and > 470 msec for females; additional ECGs may be performed if required
* Complete bundle branch blocks and other conduction abnormalities other than mild first degree atrio-ventricular block
* Irregular rhythms other than sinus arrhythmia or occasional, rare supraventricular ectopic beats
* History of unexplained syncope
* Family history of unexplained sudden death or sudden death due to long QT syndrome
* T-wave configurations are not of sufficient quality for assessing QT interval, as determined by the MI
* Show evidence of human immunodeficiency virus (HIV) and/or positive human HIV antibodies, hepatitis C and/or positive hepatitis C antibody, or hepatitis B and/or positive hepatitis B surface antigen (HBsAg)
* Intend to use over-the-counter or prescription medication within 5 days prior to dosing, other than daily multi-vitamin therapy, stable thyroid hormone replacement or medication assessed as acceptable by the MI and not interfering with the integrity of the study data collection. Medications for benign indications in healthy participants may be continued, with the exception of drugs that may alter adrenal function, blood pressure or potassium
* Have donated blood of more than 50 milliliters (mL) of blood within 60 days prior to dosing
* Have an average weekly alcohol intake that exceeds 21 units per week or participants unwilling to stop alcohol within 48 hours of entry into study until discharge each period (1 unit = 12 ounces (oz) or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits)
* Have an abnormal blood pressure (supine) defined as diastolic blood pressure >95 or less than (<) 50 millimeters of mercury (mmHg) and/or systolic blood pressure >150 or <90 mmHg confirmed by at least 1 repeat measurement
* Regularly use known drugs of abuse or show positive findings for such use on urinary drug screening
* Use of natural licorice (glycyrrhizinic acid) within 5 days of enrollment or use during the study
* Are unwilling to abstain from using grapefruit-containing products and salt-substitutes containing potassium for the duration of the study
* Have serum potassium >upper limit of normal (result from suspected hemolyzed sample may be repeated) or <lower limit of normal per lab reference range
* Have serum creatinine >124 micromoles per liter (μmol/L) (male); >106 μmol/L (female)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2013-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Clinically Significant Adverse Events (AEs) or Any Serious AEs | Baseline to 10 Days Post Dose (Estimated up to 8 Weeks)

SECONDARY OUTCOMES:
Pharmacokinetics: Maximum Serum Concentration (Cmax) of LY3045697 | Baseline to 72 Hours Post Dose
Pharmacokinetics: Area Under the Serum Concentration-Time Curve (AUC) from Zero to Infinity (AUC 0-∞) of LY3045697 | Baseline to 72 Hours Post Dose

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM-5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zuidlaren, Netherlands